CLINICAL TRIAL: NCT02091219
Title: The Effects of Vitamin D3 Versus 25OHD3 (HyD) on Serum Vitamin D Metabolites and Markers of Mineral Metabolism and Immune Function
Brief Title: Effects of Vitamin D3 Versus 25OHD3 on Mineral Metabolism and Immune Function
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, John Adams, M.D., Professor, Department of Orthopaedic Surgery, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UL1TR000124-1954; 1P50AR063020-01 (NIH); UL1TR000124 (NIH)
Record Dates: First submitted 2014-03-12; First posted 2014-03-19 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Vitamin D Deficiency
Keywords: Hypovitaminosis D; Free 25-hydroxyvitamin D; Total 25-hydroxyvitamin D
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Vitamin D; Cholecalciferol; Calcifediol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 25(OH)D3 (Experimental): 20 micrograms/day by mouth for 16 weeks
  Interventions: Drug: 25(OH)D3
- Vitamin D3 (Experimental): 2,400 IU/day by mouth for 16 weeks
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D — 2400 IU/day by mouth for 16 weeks
  Other Names: Cholecalciferol
  Arms: Vitamin D3
Drug: 25(OH)D3 — 20 micrograms/day by mouth for 16 weeks
  Other Names: Calcifediol; HyD
  Arms: 25(OH)D3

SUMMARY:
The purpose of this study is to compare the effects of two different forms of vitamin D supplements (vitamin D3 and 25-hyrdroxyvitamin D3 [25(OH)D3]) on vitamin D levels in the blood, and on markers of skeletal and immune health. This study is designed as a pilot study. A multi-ethnic cohort of 48 patients will be included (12 Caucasian, 12 African American, 12 Hispanic/Latino, 12 Asian/Asian American). Potential study candidates will undergo a screening visit during which a medical history will be taken, a physical exam performed, a dietary questionnaire administered, and blood collected. The purpose of the screening visit is to identify vitamin D-deficient (25-hydroxyvitamin D <20 ng/ml) individuals who are candidates for vitamin D supplementation. Eligible patients will then be randomly assigned to receive either vitamin D3 (2400 IU/day) or 25(OH)D3 (20 mcg/day) for 16 weeks. After initiating supplementation, study patients will return for follow-up visits at weeks 4, 8, and 16. At each visit, blood will be collected to assess vitamin D levels in the blood, as well as markers of skeletal and immune function. Participation in this study will therefore involve a total of 5 visits (1 screening visit, 1 randomization visit during which participants will receive their study supplements, 3 follow-up visits). After all data is collected, changes in vitamin D levels in the blood following supplementation with either vitamin D3 versus 25(OH)D3 will be determined, and correlated to markers of calcium balance and immune function. Knowledge gained from this study may have a significant impact on how vitamin D status is defined, and how vitamin D repletion is administered.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* 25D < 20 mg/ml

Exclusion Criteria:

* Age < 18
* 25D > 20 ng/ml at time of screening
* Clear signs of infection at time of screening (coughing, sneezing, wheezing, frequency, dysuria)
* History of conditions that would influence intestinal absorption of vitamin D3 or 25OHD3 supplements
* History of nephrolithiasis, primary hyperparathyroidism, or other metabolic bone disease
* History of chronic kidney disease (defined as CrCl < 30 ml/min)
* History of rheumatologic or autoimmune conditions
* History of sarcoidosis
* History of active or latent tuberculosis
* History of HIV
* History of hyperthyroidism
* History of chronic glucocorticoid use defined as the equivalent of 5 mg of prednisone per day for more than 2 months within the last 6 months
* History of use of medications known to affect calcium/vitamin D metabolism, bone metabolism, and immune response
* Hypercalcemia
* Hypercalcinuria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-06; Primary Completion 2019-12 (Actual); Study Completion 2019-12-07 (Actual)

PRIMARY OUTCOMES:
Change in total serum 25D | 16 weeks

SECONDARY OUTCOMES:
Change in serum free 25D | 16 weeks
Change in serum total 1,25D | 16 weeks
Change in total free 1,25D | 16 weeks
Change in serum calcium | 16 weeks
Change in urinary calcium | 16 weeks
Change in serum iPTH | 16 weeks
Change in serum bone turnover markers | 16 weeks
Change in markers of immune function | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John S Adams, MD, Principal Investigator — University of California, Los Angeles Department of Orhtopaedic Surgery
Locations (2):
- United States (2):
  - UCLA Clinical and Translational Research Center (CTRC), Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California

REFERENCES:
- [Derived] Shieh A, Lee SM, Lagishetty V, Gottleib C, Jacobs JP, Adams JS. Pilot Trial of Vitamin D3 and Calcifediol in Healthy Vitamin D Deficient Adults: Does It Change the Fecal Microbiome? J Clin Endocrinol Metab. 2021 Nov 19;106(12):3464-3476. doi: 10.1210/clinem/dgab573. PMID 34343292
- [Derived] Shieh A, Ma C, Chun RF, Wittwer-Schegg J, Swinkels L, Huijs T, Wang J, Donangelo I, Hewison M, Adams JS. Associations Between Change in Total and Free 25-Hydroxyvitamin D With 24,25-Dihydroxyvitamin D and Parathyroid Hormone. J Clin Endocrinol Metab. 2018 Sep 1;103(9):3368-3375. doi: 10.1210/jc.2018-00515. PMID 29931358